CLINICAL TRIAL: NCT03488186
Title: A Randomized, Open Label, Parallel, Single and Multiple Doses Designed Clinical Study to Evaluate Comparative Pharmacokinetics (PK)-Pharmacodynamics (PD) After Oral Administration of Lansoprazole Capsules and Lansoprazole Enteric-coated Capsules in Healthy Chinese Volunteers
Brief Title: PK-PD Comparative Study of Lansoprazole Capsules and Lansoprazole Enteric-coated Capsules in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Beijing Xuze Medical Technology Co., LTD. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC00-018-02
Record Dates: First submitted 2018-03-18; First posted 2018-04-04 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Effect of Drugs; Safety Issues
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lansoprazole Capsules (Experimental): Lansoprazole Capsules of Beijing Sihuan Pharm, 30 mg
  Interventions: Drug: Lansoprazole Capsules
- Lansoprazole enteric-coated Capsules (Active Comparator): Lansoprazole enteric-coated Capsules of Takeda Pharmaceutical Company Limited, 30 mg
  Interventions: Drug: Lansoprazole Capsules

INTERVENTIONS:
Drug: Lansoprazole Capsules — 24 healthy volunteers will be recruited and randomized into 2 groups (12 for each). During the study session, subjects will receive T drug in group A or R drug in group B for 7 days in fasted condition.

SUMMARY:
The objective of this study was to compare the relative PK-PD of Lansoprazole Capsules and Lansoprazole DR Capsules in healthy Chinese volunteers.

DETAILED DESCRIPTION:
This is a randomized, open Label, parallel, single and multiple doses designed clinical trial. This study will determine the pharmacokinetics (PK), pharmacodynaimcs (PD) and safety after oral administration of an investigational Lansoprazole Capsules in healthy Chinese volunteers.

This study will enroll 24 healthy adults with 12 cases in each group (male : female=1:1).

ELIGIBILITY:
Inclusion Criteria:

* Subject who were healthy, adult, human beings within 18 and 60 years of age (both inclusive).
* Male (weight ≥50kg) or female (weight ≥45kg); Subject having a body mass index between 19.0 and 26.0 (both inclusive), calculated as weight in Kg/height in m2.
* Subject who totally understand the aim, procedure, benefits and adverse effects of this clinical trial, make decision by his/her free will, and sign a consent form to follow the progress;
* The participant could communicate well with investigator, comply with and finish the study according to the procedure.

Exclusion Criteria:

* Subject who has past or present history of any serious diseases, including (but not limited to) digestive, cardiovascular, respiratory, urinary, musculoskeletal, endocrine, psychiatric or neurological, hematologic, immunological or metabolic disorders;
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator;
* Intake of over the counter (OTC) or prescribed medications or vitamins or any traditional medicine products for the last 14 days before first dosing.
* Has a special requirement for food and cannot adhere to a uniform diet or swallowing victims.
* Cannot tolerate placement of the pH probe;
* Venous puncture intolerable and/or blood phobia
* Abused of tea, coffee and caffeine-contained beverages; or taking caffeine/xanthene containing food or beverages (like tea, coffee, chocolates and cola drinks) for the last 48 hrs before first dosing.
* Habit of alcoholism; or frequent drinkers for the last 6 months before screening; or intake of any alcoholic products for the last 24 hrs before first dosing.
* Regular smoker who has a habit of smoking more than five cigarettes per day for the last 3 months and has difficulty in abstaining from smoking during sample collection period.
* Blood donation or blood loss ≥ 450 mL for the last 3 months before first dosing; or plan to donate blood or blood composition during the study or 3 months after the end of the study.
* Intake of any enzyme modifying food or beverages for the last 48 hrs before first dosing.
* Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study; or subjects declined to practice non-pharmacologic prevention of birth control during the study.
* Abused of drugs or Intake of drugs for the last 3 months before screening.
* Subjects who had participated in any other clinical investigation using experimental drug/medical instrument/diagnostic reagent in past 3 months before screening.
* Clinically significant abnormalities judged by investigators during screening test.
* Positive breath test result for H pylori at Screening;
* Confirmed positive in alcohol screening, smoking screening or selected drug of abuse.
* Human immunodeficiency virus(HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or syphilis positive.
* Other reasons for non-inclusion judged by investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Assessment | 16 hrs post-dose on day 1 and day 7.
  1. Cmax: Maximum Observed Plasma Concentration for lansoprazole Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
     [Time Frame: 16 hours post-dose on Day 1 and D7]
  2. TmaxTime to Reach the Maximum Plasma Concentration [Time Frame: 16 hours post-dose on Day 1 and D7]
  3. AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for lansoprazole AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity [Time Frame: Time Frame: 16 hours post-dose on Day 1 and D7] model.
PD Assesment | 24 hrs post-dose on day 1 and day 7.
  1. Percentage time with the intragastric potential of hydrogen (pH)<4 Duration of intragastric pH<4 within 24 hours postdose
  2. Percentage time with the intragastric pH>6 Duration of intragastric pH>6 within 24 hours postdose
  3. The time of the intragastric pH reaching 4The time of intragastric pH reaching 4 after the last dos
  4. The time of the intragastric pH reaching 6The time of intragastric pH reaching 6 after the last dose

SECONDARY OUTCOMES:
Duration of intragastric pH within 24 hours postdose | 24 hrs after dose on day 1 and 7
  ean intragastric pH per hour Mean intragastric pH per hour Percentage time with the intragastric pH>4 during the first 4 hours Duration of intragastric pH>4 within first 4 hours postdose Percentage time with the intragastric pH>6 during the first 4 hours Duration of intragastric pH>6 within first 4 hours postdose Percentage of the participants with duration time of intragastric pH>4 over 12hNumbers of participants with duration time of intragastric pH>4 over 16h Percentage of the participants with duration time of intragastric pH>6 over 12h Numbers of participants with duration time of intragastric pH>6 over 16h intragastric pH<4 within 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Wu, Doctor, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No